CLINICAL TRIAL: NCT06423573
Title: A Long-term Non-interventional Study to Assess the Incidence of Skin Malignancies in Patients With Dystrophic and Junctional Epidermolysis Bullosa Receiving Treatment With Filsuvez
Brief Title: A Study to Assess the Incidence of Skin Cancers in Patients With Epidermolysis Bullosa Receiving Filsuvez
Acronym: FOSteR
Status: Recruiting | Type: Observational
Sponsor: Amryt Pharma (Industry)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: AEB-21
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Epidermolysis Bullosa, Dystrophic; Epidermolysis Bullosa, Junctional
Keywords: Filsuvez; Birch bark extract
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa, Junctional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with dystrophic or junctional EB being treated with Filsuvez: Patients in this cohort will be receiving treatment with Filsuvez for their EB.
  Interventions: Drug: Filsuvez
- Patients with dystrophic or junctional EB not being treated with Filsuvez: Patients in this cohort will be receiving treatment other than Filsuvez or no treatment at all for their EB.

INTERVENTIONS:
Drug: Filsuvez — Topical gel
  Other Names: Birch bark extract
  Groups: Patients with dystrophic or junctional EB being treated with Filsuvez

SUMMARY:
In patients with epidermolysis bullosa (EB), collagen does not form properly, so their skin is very fragile and blisters easily. Such patients are also at greatly increased risk of developing skin cancers. Filsuvez is a topical gel used to promote healing of skin lesions in patients with certain types of EB. In this observational study, patients with either dystrophic EB (DEB) or junctional EB (JEB) will receive standard of care treatment, whether Filsuvez or something else, and will be followed for up to 5 years. The main purpose is to see if the use of Filsuvez affects the likelihood of developing skin malignancies in these patient populations.

DETAILED DESCRIPTION:
Some forms of EB are associated with a greatly increased incidence of aggressive skin and mucosal squamous cell carcinoma (SCC), as well as increased incidence of other skin malignancies including basal cell carcinoma (BCC) and malignant melanoma (MM). This long-term non-interventional study will assess all types of skin malignancies (SCC, BCC, and MM) in DEB and JEB patients. It is an observational study of real-world treatment practices, in which patients will receive standard of care therapy whatever that may entail. Data will be obtained from two sources: clinical study centers in the European Union (EU) and the United Kingdom (UK), and pre-existing EB registries in the EU. Participants will be followed for up to 5 years, and information about the development and nature of skin malignancies will be collected over this time period both from patients who are taking and those who are not taking Filsuvez.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of dystrophic EB or junctional EB

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with dystrophic EB or junctional EB, whether they are receiving Filsuvez, receiving another treatment for EB, or not receiving any treatment.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2031-11-30 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of first skin malignancy during follow-up in EB patients receiving Filsuvez | Up to 5 years
  Patients being treated with Filsuvez will be followed for occurrence of skin malignancies from the date of study enrolment until either the date of discontinuation (withdrawal of consent, withdrawal from the site or registry, physician decision, death, or lost to follow-up) or termination of the study

SECONDARY OUTCOMES:
Incidence of first skin malignancy during follow-up in EB patients not receiving Filsuvez | Up to 5 years
  Patients with EB who are not being treated with Filsuvez will be followed for occurrence of skin malignancies from the date of study enrolment until either the date of discontinuation (withdrawal of consent, withdrawal from the site or registry, physician decision, death, or lost to follow-up) or termination of the study

CONTACTS AND LOCATIONS:
Locations (5):
- CHU de Toulouse, Hôpital Larrey, Toulouse, France
- Hospital of Skin and Venereal Diseases of Thessaloniki, Thessaloniki, Greece
- Spain (2):
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital San Juan de Dios (Barcelona), Barcelona
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom